CLINICAL TRIAL: NCT04496206
Title: Musculoskeletal Problems During Pregnancy
Status: Completed | Type: Observational
Sponsor: Eskisehir City Hospital (Other)
Responsible Party: Principal Investigator, Fulya Bakılan, Physical Therapy and Rehabilitation Specialist, Eskisehir City Hospital
Other Study IDs: EskisehirCityHospital
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Most Common Musculoskeletal Problems in Pregnancy
Keywords: carpal tunnel syndrome; low back pain; pelvic girdle pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Low Back Pain; Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention, it is retrospective study.

SUMMARY:
Aim: This study was conducted to identify the most common musculoskeletal problems according to trimester, experienced by pregnant women.

Material and Methods: A total of 120 pregnant women who admitted to physical medicine and rehabilitation clinic, evaluated retrospectively in this study. Application complaints, the diagnosis and the trimester of the pregnant women and also age, weight, height, number of pregnancy, working status, presence of secondary disease were recorded.

ELIGIBILITY:
Inclusion Criteria:

Pregnant patients who have age, weight, size, employment status, duration of pregnancy, nulli/multi-parity, presence of other disorders, application complaints, the diagnosis information were included to the study

Exclusion Criteria:

Non-pregnant patients and pregnant patients with missing data were excluded from the study

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: One hundred and twenty pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Application complaints | 1 day
  such as pain, numbness, tingling, swelling and cramps…
the diagnosis | 1 day
  low back pain, pelvic girdle pain, carpal tunnel syndrome, pedal edema, cramp, knee pain, foot pain, neck pain…

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakılan, Principal Investigator — Eskisehir City Hospital
Locations (1):
- Eskişehir City Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
One year later, after being published in a joournal, study information can be share with other researchers